CLINICAL TRIAL: NCT01237808
Title: Study of Low-Dose Cytarabine and Etoposide With or Without All-Trans Retinoic Acid in Older Patients Not Eligible for Intensive Chemotherapy With Acute Myeloid Leukemia and NPM1 Mutation
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Ulm (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Prof. Dr. Hartmut Doehner, Prof. Dr., University of Ulm
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AMLSG 15-10
Record Dates: First submitted 2010-11-09; First posted 2010-11-10 (Estimated); Last update posted 2018-08-01 (Actual); Status verified 2018-07

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: AML; NPM1 Mutation; elderly patients (>60 years); unfit for intensive chemotherapy
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Cytarabine; Etoposide; Tretinoin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standard arm (Active Comparator): 6 cycles of chemotherapy (low-dose cytarabine and etoposide) without ATRA
  Interventions: Drug: Cytarabine; Drug: Etoposide
- Investigational arm (Experimental): 6 cycles of chemotherapy (low-dose cytarabine and etoposide) with ATRA (All-trans-Retinoic acid)
  Interventions: Drug: Cytarabine; Drug: Etoposide; Drug: All-trans retinoic acid (ATRA)

INTERVENTIONS:
Drug: Cytarabine — in all treatment cycles: Cytarabine 20 mg/day, s.c., bid, days 1-7; (total dose 280 mg).
Drug: Etoposide — first treatment cycle Etoposide 50 mg/m²/day, continuously i.v., days 1-3; (total dose 150 mg/m2) treatment cycles 2 to 6 Etoposide 100 mg/day, p.o. or i.v. (over 1 hour), days 1-3; (total dose 300 mg).
Drug: All-trans retinoic acid (ATRA) — in all treatment cycles: ATRA 45 mg/m²/day p.o., days 8-10, ATRA 15 mg/m²/day p.o., days 11-28, with or shortly after meals distributed on 3 doses per day.
  Arms: Investigational arm

SUMMARY:
This is a randomized, Phase-III, two-arm, open-label, multi-center study in adult patients with AML and NPM1 mutation ineligible for intensive chemotherapy.

Sample size: 144 patients

Investigator's sites: 50-55 sites in Germany and Austria (2-10 patients per trial site are expected to be included into the trial)

Estimated treatment duration of an individual patient: 8 months (Follow-Up period per patient will last additional 2 years)

ELIGIBILITY:
Inclusion Criteria:

* Patients with confirmed diagnosis of acute myeloid leukemia according to the World Health Organization (WHO) classification (including de novo AML, t-AML and s-AML)
* Presence of NPM1 mutation as assessed in one of the central AMLSG reference laboratories.
* Age > 60 years. There is no upper age limit.
* No prior chemotherapy for leukemia except hydroxyurea to control hyperleukocytosis if needed for up to 10 days during the diagnostic screening phase.
* Signed written informed consent
* Men must give their informed consent that they do not father a baby and must use a latex condom during any sexual contact with women of childbearing potential, even if they have undergone a successful vasectomy. (while on therapy and for 3 month after the last dose of chemotherapy)
* WHO performance status ≤ 3
* Patients not eligible for intensive chemotherapy according to at least one of the following criteria

  * HCT-CI Score >2
  * Patient's decision
  * age ≥ 75 years

Exclusion Criteria:

The presence of any of the following will exclude a patient from study enrollment:

* All other AML subtypes, in particular those AML with other recurrent genetic changes (according to WHO 2008):

  * AML with t(8;21)(q22;q22); RUNX1-RUNX1T1
  * AML with inv(16)(p13.1q22) or t(16;16)(p13.1;q22); CBFB-MYH11
  * AML with t(15;17)(q22;q12); PML-RARA (or other translocations involving RARA)
  * AML with t(9;11)(p22;q23); MLLT3-MLL (or other translocations involving MLL)
  * AML with t(6;9)(p23;q34); DEK-NUP214
  * AML with inv(3)(q21q26.2) or t(3;3)(q21;q26.2); RPN1-EVI1
* No consent for registration, storage and processing of the individual disease-characteristics and course as well as information of the family physician and all other treating physicians about study participation
* Bleeding disorder independent of leukemia
* Uncontrolled infection
* Known positive for HIV, HBV or HCV
* Organ insufficiency (creatinine >1.5x upper normal serum level; bilirubin, AST or ALP >2.5x upper normal serum level, not attributable to AML; heart failure NYHA III/IV; severe obstructive or restrictive ventilation disorder)
* Severe neurological or psychiatric disorder interfering with ability of giving an informed consent
* Patients with a "currently active" second malignancy other than non-melanoma skin cancers. Patients are not considered to have a "currently active" malignancy if they have completed therapy and are considered by their physician to be at less than 30% risk of relapse within one year.

Min Age: 61 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2011-03; Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
overall survival | 2 years and 8 months

SECONDARY OUTCOMES:
Rate of Complete remission | 8 months
cumulative incidence of relapse | 2 years and 8 months
cumulative incidence of death in complete remission | 2 years and 8 months
event-free survival | 2 years and 8 months
Rate of early deaths (ED)/hypoplastic deaths (HD) | 8 months
Type, frequency, severity, timing and relatedness of adverse events (AEs) and laboratory abnormalities observed during different treatment cycles | 8 months
  adverse events graded using the National Cancer Institute Common Terminology Criteria for Adverse Events [NCI CTCAE] Version 4.0
Incidence of infection after each treatment cycle | 8 months
Duration of neutropenia after each treatment cycle | 8 months
Duration of thrombocytopenia after each treatment cycle | 8 months
Duration of hospitalization after each treatment cycle | 8 months
Quality of life | 2 years and 8 months
  assessed by the EORTC Quality of Life Core Questionnaire (QLQ-C30), supplemented by information on self-assessed concomitant diseases, late treatment effects, and demographics according to Messerer et al.33

CONTACTS AND LOCATIONS:
Overall Officials: Hartmut Döhner, MD, Principal Investigator — University Hospital of Ulm
Locations (33):
- Germany (33):
  - Ubbo-Emmius Klinik Aurich, Aurich
  - Charité Universitätsmedizin Berlin, Berlin
  - University Hospital of Bonn, Bonn
  - Städtisches Klinikum Braunschweig, Braunschweig
  - Klinikum Bremen-Mitte gGmbH, Bremen
  - Kliniken Essen Süd, Evangelischs Krankenhaus, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Medizinische Universitätsklinik, Freiburg im Breisgau
  - Medizinisches Versorgungszentrum Osthessen GmbH, Fulda
  - Universitätsklinikum Gießen, Giessen
  - Wilhelm- Anton- Hospital gGmbH, Goch
  - Universitätsmedizin Göttingen, Göttingen
  - University Hospital of Hamburg Eppendorf, Hamburg
  - Asklepios Klinik Altona, Hamburg
  - Medical Department III, Hospital of Hannover-Siloah, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - SLK-Kliniken Heilbronn GmbH, Heilbronn
  - Department of Internal Medicine I, University Hospital of Saarland, Homburg
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
  - Department of Interial Medicine /Hematology and Oncology, Caritas Hospital Lebach, Lebach
  - Klinikum der Johannes Gutenberg Universität Mainz, Mainz
  - Stauferklinikum Schwäbisch Gmünd, Mutlangen
  - Klinikum rechts der Isar der TU Muenchen, München
  - Pius Hospital Oldenburg, Oldenburg
  - Krankenhaus der Barmherzigen Brueder, Regensburg
  - Caritas-Klinik St. Theresia, Saarbrücken
  - Clinikal Cetner of Stuttgart, Center of Oncology, Stuttgart
  - Diakonie-Klinikum Stuttgart, Stuttgart
  - Krankenhaus der Barmherzigen Brüder Trier, Trier
  - Universitätsklinikum Tübingen, Tübingen
  - University hospital of Ulm, Ulm
  - Medical Center II - Hematology/Oncology, Clinical Center Villingen-Schwenningen, Villingen-Schwenningen
  - Helios Klinikum Wuppertal, Wuppertal